CLINICAL TRIAL: NCT03433508
Title: Restrictive Versus Liberal Red Blood Cell Transfusion in Patients of Cirrhosis With Septic Shock: An Open Label Randomized Controlled Trial
Brief Title: Restrictive Versus Liberal Red Blood Cell Transfusion in Patients of Cirrhosis With Septic Shock
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-cirrhosis-01
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal (Experimental): 2 PRBC /day to maintain the target of Hemoglobin 10 to 11 gm/dL. PRBC will be given intravenously at least for 28 days
  Interventions: Biological: Liberal
- Restrictive (Active Comparator): To maintain the target Hemoglobin of 7 to 8 gm/dL.
  Interventions: Other: Restrictive

INTERVENTIONS:
Biological: Liberal — 2 PRBC /day to maintain the target of Hemoglobin 10 to 11 gm/dL. PRBC will be given intravenously at least for 28 days
  Arms: Liberal
Other: Restrictive — To maintain the target Hemoglobin of 7 to 8 gm/dL.
  Arms: Restrictive

SUMMARY:
Consecutive cirrhotics who present to emergency department of ILBS with documented or suspected sepsis induced hypotension with Hb <8 gm/dl will be randomly assigned to restrictive (Target Hb 7-8 gm/dl) to liberal (Target Hb 10-11 gm/dl) group in a 1:1 proportion At admission, all patients will undergo physical examination and baseline investigations to identify site of sepsis. Enrolled patients will be given PRBC-transfusion (Not more than two units of PRBC/day) when they reach their assigned trigger value (Hb 7-8 g/dl or 10-11 g/dl ) during the entire ICU stay. All other interventions will be at the discretion of clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis with septic shock.
2. Age >18 years

Exclusion Criteria:

1. Previous severe adverse reaction with blood products,
2. Disseminated intravascular coagulopathy
3. HCC
4. Pregnancy
5. Malignancy
6. Active gastrointestinal bleeding
7. Intracranial bleeding
8. Chronic Kidney disease with Maintenance Hemodialysis
9. Pulmonary Edema
10. Congestive Heart Failure
11. Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Mortality in both groups | 28 dyas

SECONDARY OUTCOMES:
Improvement in vasopressors in both groups | 28 days
  Improvement is defined as tapering the dose of vasopressors
Incidence of complications in both groups | 28 days
Length of ICU (Intensive Care Unit) stay | 28 days
Requirement of mechanical ventilation in both groups | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided